CLINICAL TRIAL: NCT01769404
Title: Evaluation of the Counter-Regulatory Response to Hypoglycaemia Following LY2605541 Administration Compared to Insulin Glargine in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of LY2605541 and Glargine in Participants With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 14870; I2R-MC-BIDM (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2019-06-24 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-03

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2605541 (Experimental): Stable dose of LY2605541 (0.2 to 0.6 units per kilogram [U/kg]) administered subcutaneously (SQ) once daily for at least 14 days in 1 of 2 treatment periods. Dose based on prestudy basal insulin dosing regimen.
  Interventions: Biological: LY2605541
- Insulin Glargine (Active Comparator): Stable dose of insulin glargine (0.2 to 0.6 U/kg) administered SQ once daily for at least 14 days in 1 of 2 treatment periods. Dose based on prestudy basal insulin dosing regimen.
  Interventions: Biological: Insulin Glargine

INTERVENTIONS:
Biological: LY2605541
  Arms: LY2605541
Biological: Insulin Glargine
  Arms: Insulin Glargine

SUMMARY:
This study has 2 parts. Each participant will receive a daily injection of LY2605541 during one treatment period and a daily injection of insulin glargine during one treatment period. Each treatment period is 2 to 3 weeks and is followed by a procedure to lower blood sugar levels to see how the body recovers after each treatment.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetic for more than 1 year with glycated hemoglobin (HbA1c) less than 9%
* Otherwise fit and healthy
* Nonsmoker

Exclusion Criteria:

* Taking medication or supplements other than insulin to control diabetes
* Suffered a hypoglycemic event in the last 12 months that required hospitalization or has poor awareness of hypoglycemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Neuss, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.
Groups:
- Cohort 1 (LY2605541, Then Insulin Glargine): Participants received a stable dose of 0.2 to 0.6 U/kg LY2605541, administered subcutaneously (SQ), once daily for 14 days in Treatment Period 1, followed by a stable dose of 0.2 to 0.6 U/kg insulin glargine, administered SQ, once daily for 14 days in Treatment Period 2.
- Cohort 2 (Insulin Glargine, Then LY2605541): Participants received a stable dose of 0.2 to 0.6 U/kg insulin glargine, administered SQ, once daily for 14 days in Treatment Period 1, followed by a stable dose of 0.2 to 0.6 U/kg LY2605541, administered SQ, once daily for 14 days in Treatment Period 2.
Period: Treatment Period 1
Arm/Group | Cohort 1 (LY2605541, Then Insulin Glargine) | Cohort 2 (Insulin Glargine, Then LY2605541)
Started | 12 | 13
Received at Least 1 Dose of Study Drug | 9 | 13
Completed | 7 | 13
Not Completed | 5 | 0
Not completed — Did not meet eligibility criteria | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Sponsor decision | 1 | 0
Period: Treatment Period 2
Arm/Group | Cohort 1 (LY2605541, Then Insulin Glargine) | Cohort 2 (Insulin Glargine, Then LY2605541)
Started | 7 | 13
Completed | 0 | 13
Not Completed | 7 | 0
Not completed — Sponsor decision | 7 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- All Participants: All participants who received at least 1 dose of study drug.
Arm/Group | All Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 22

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Epinephrine
Description: Epinephrine levels are presented. Each participant's measurements at 30, 15, and 0 minutes preclamp on the day of the clamp were averaged for the baseline value, and measurements at blood glucose (BG) level attainment and +10, 20, and 30 minutes were averaged for the BG nadir value.
Time Frame: 30, 15, and 0 minutes Preclamp; 10, 20, and 30 minutes Post-Clamp
Population: All participants in Cohort 2 who received at least 1 dose of study drug with evaluable epinephrine data. As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: picomole per liter (pmol/L)
Groups:
- LY2605541: Participants received a stable dose of LY2605541 (0.2 to 0.6 U/kg) administered SQ once daily for at least 14 days. Dose based on prestudy basal insulin dosing regimen.
- Insulin Glargine: Participants received a stable dose of insulin glargine (0.2 to 0.6 U/kg) administered SQ once daily for at least 14 days. Dose based on prestudy basal insulin dosing regimen.
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 13 | 13
picomole per liter (pmol/L)
  Baseline | 157.2 (90.9) | 196.5 (207.0)
  BG nadir | 607.5 (281.0) | 525.2 (305.4)

2. Secondary Outcome: Amount of Glucose Required to Reach Blood Glucose (BG) of 72 mg/dL
Description: The amount of infused glucose required to reach BG of 72 milligrams per deciliter (mg/dL) is presented.
Time Frame: 30, 15, and 0 minutes Preclamp; 10, 20, and 30 minutes Post-Clamp
Population: All participants in Cohort 2 who received at least 1 dose of study drug with evaluable BG data. As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams (mg)
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 13 | 13
milligrams (mg) | 11600 (37) | 12700 (43)

3. Secondary Outcome: Amount of Glucose Required to Maintain BG of 72 mg/dL
Description: The amount of infused glucose required to maintain BG of 72 mg/dL for 1 hour is presented.
Time Frame: 30, 15, and 0 minutes Preclamp; 10, 20, and 30 minutes Post-Clamp
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 13 | 13
mg | 15400 (34) | 15900 (37)

4. Secondary Outcome: Concentration of Cortisol
Description: Cortisol levels are presented. Each participant's measurements at 30, 15, and 0 minutes preclamp on the day of the clamp were averaged for the baseline value, and measurements at BG level attainment and +30 minutes were averaged for the BG nadir value.
Time Frame: 30, 15, and 0 minutes Preclamp; 10, 20, and 30 minutes Post-Clamp
Population: All participants in Cohort 2 who received at least 1 dose of study drug with evaluable cortisol data. As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: nanomole per liter (nmol/L)
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 13 | 13
nanomole per liter (nmol/L)
  Baseline | 206.7 (75.4) | 260.0 (92.4)
  BG nadir | 337.3 (121.2) | 333.8 (74.0)

5. Secondary Outcome: Concentration of Glucagon
Description: Glucagon levels are presented. Each participant's measurements at 30, 15, and 0 minutes preclamp on the day of the clamp were averaged for the baseline value, and measurements at BG level attainment and +30 minutes were averaged for the BG nadir value.
Time Frame: 30, 15, and 0 minutes Preclamp; 10, 20, and 30 minutes Post-Clamp
Population: All participants in Cohort 2 who received at least 1 dose of study drug with evaluable glucagon data. As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 13 | 13
pmol/L
  Baseline | 8.02 (2.88) | 5.28 (2.46)
  BG nadir | 5.89 (2.82) | 4.98 (2.79)

6. Secondary Outcome: Concentration of Growth Hormone
Description: Growth hormone levels are presented. Each participant's measurements at 30, 15, and 0 minutes preclamp on the day of the clamp were averaged for the baseline value, and measurements at BG level attainment and +30 minutes were averaged for the BG nadir value.
Time Frame: 30, 15, and 0 minutes Preclamp; 10, 20, and 30 minutes Post-Clamp
Population: All participants in Cohort 2 who received at least 1 dose of study drug with evaluable growth hormone data. As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: micrograms per liter (µg/L)
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 13 | 13
micrograms per liter (µg/L)
  Baseline | 1.0816 (2.5527) | 1.3948 (1.3981)
  BG nadir | 6.8752 (6.7187) | 8.0114 (9.9621)

7. Secondary Outcome: Concentration of Norepinephrine
Description: Norepinephrine values are presented. Each participant's measurements at 30, 15, and 0 minutes preclamp on the day of the clamp were averaged for the baseline value, and measurements at BG level attainment and +10, 20, and 30 minutes were averaged for the BG nadir value.
Time Frame: 30, 15, and 0 minutes Preclamp; 10, 20, and 30 minutes Post-Clamp
Population: All participants in Cohort 2 who received at least 1 dose of study drug with evaluable norepinephrine data. As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | LY2605541 | Insulin Glargine
Number analyzed (Participants) | 13 | 13
pmol/L
  Baseline | 1004.2 (358.2) | 1139.8 (603.2)
  BG nadir | 1235.8 (422.8) | 1434.8 (933.3)

ADVERSE EVENTS:
Groups:
- Cohort 1: 0.2-0.6 U/kg LY2605541; Cohort 2: 0.2-0.6 U/kg LY2605541: Participants received a stable dose of LY2605541 (0.2 to 0.6 U/kg) administered SQ once daily for at least 14 days in Treatment Period 1 or 2. Dose based on prestudy basal insulin dosing regimen.
- Cohort 1: 0.2-0.6 U/kg Insulin Glargine; Cohort 2: 0.2-0.6 U/kg Insulin Glargine: Participants received a stable dose of insulin glargine (0.2 to 0.6 U/kg) administered SQ once daily for at least 14 days in Treatment Period 1 or 2. Dose based on prestudy basal insulin dosing regimen.
Arm/Group | Cohort 1: 0.2-0.6 U/kg LY2605541 | Cohort 1: 0.2-0.6 U/kg Insulin Glargine | Cohort 2: 0.2-0.6 U/kg LY2605541 | Cohort 2: 0.2-0.6 U/kg Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 1/9 | 3/7 | 1/13 | 3/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: 0.2-0.6 U/kg LY2605541 (N=9) | Cohort 1: 0.2-0.6 U/kg Insulin Glargine (N=7) | Cohort 2: 0.2-0.6 U/kg LY2605541 (N=13) | Cohort 2: 0.2-0.6 U/kg Insulin Glargine (N=13)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
As per protocol amendment, no participants in cohort 1 were analyzed and only cohort 2 participants were analyzed for efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days